CLINICAL TRIAL: NCT05572996
Title: Inhaled Treprostinil Expanded Access Program in Pulmonary Hypertension Associated With Interstitial Lung Disease
Status: Available | Type: Expanded Access
Sponsor: Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: FITREP-EAP2201
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Pulmonary Hypertension; Interstitial Lung Disease; Combined Pulmonary Fibrosis and Emphysema
Keywords: Inhaled Treprostinil; Tyvaso; EAP; Expanded Access; Early Access; Compassionate Use; Named Patient Program; NPP; PH-ILD
MeSH Terms: conditions — Hypertension, Pulmonary; Lung Diseases, Interstitial; Emphysema | interventions — treprostinil

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Inhaled Treprostinil
  Other Names: Tyvaso

SUMMARY:
This is an Expanded Access Program (EAP) for eligible participants with Pulmonary Hypertension associated with Interstitial Lung Disease (PH-ILD) designed to provide access to Inhaled Treprostinil. Availability will depend on territory elegibility.

ELIGIBILITY:
Inclusion Criteria:

1. Patient consent
2. Males and females aged 18 years old or older
3. PH-ILD diagnosis:

   * Confirmed diagnosis of Group 3 PH by Right Heart Catheterization (RHC):

     - mPAP > 20 mmHg with PAWP ≤ 15 mmHg and PVR ≥ 2 WU and
   * Confirmed diagnosis of diffuse parenchymal lung disease based on imaging (any form of ILD or CPFE)

Exclusion Criteria:

1. Diagnosis of PAH or PH for reasons other than Group 3 PH-ILD
2. Use of concomitant PAH drugs contraindicated for PH-ILD (ambrisentan and riociguat)
3. Use of any concomitant investigational drug

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult